CLINICAL TRIAL: NCT01414166
Title: A 16-Week, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Extended Release Niacin/Laropiprant in South and Southeast Asians Not on a Lipid Modulating Agent, With Decreased High-Density Lipoprotein Cholesterol and Low- Density Lipoprotein Cholesterol at or Below NCEP ATP III Goal
Brief Title: Niacin/Laropiprant Tablet for South and Southeast Asians With Low High-Density Lipoprotein Cholesterol (LDL-C) at Risk for Cardiovascular Disease (MK-0524A-108)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In HPS2-THRIVE, MK-0524A did not meet the primary efficacy objective and there was a significant increase in incidence of some types of non-fatal SAEs
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0524A-108; CTRI/2012/08/002873 (Registry Identifier: CTRI)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERN/LRPT group (Experimental): All participants will begin with a screening period of 1 week, followed by a placebo run-in period of 2 weeks before being randomized to receive ERN/LRPT for 16 weeks.
  Interventions: Drug: ERN/LRPT
- Placebo group (Placebo Comparator): All participants will begin with a screening period of 1 week, followed by a placebo run-in period of 2 weeks before being randomized to receive placebo for 16 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ERN/LRPT — ERN/LRPT combination tablets (each containing 1 g of extended release niacin and 20 mg of laropiprant), orally, one tablet once per day for 4 weeks, then 2 tablets once per day for 12 weeks
  Other Names: Tredaptive™
  Arms: ERN/LRPT group
Drug: placebo — ERN/LRPT-matched placebo, orally, one tablet once per day for 4 weeks, then 2 tablets once per day for 12 weeks
  Arms: Placebo group

SUMMARY:
The study will evaluate the use of extended release niacin/laropiprant (ERN/LRPT) combination tablets in a primary prevention population currently not taking or eligible for lipid-modifying therapy (LMT); the population will comprise participants with low to moderate risk for coronary heart disease (CHD), low high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C) at or below goal level, and normal or mildly elevated triglyceride (TG) levels.

ELIGIBILITY:
Inclusion criteria:

* LMT ineligible
* Participants must meet the lipid criteria of "low to moderate CHD risk" as defined by National Cholesterol Education Program Adult Treatment Panel III Framingham Point Scores (NCEP ATP III)
* HDL-C <40 mg/dL (1.03 mmol/L) in males and <50 mg/dL (1.29 mmol/L) in females
* Triglyceride (TG) level <300 mg/dL (3.39 mmol/L).
* Fasting serum glucose (FSG) at Visit 1 AND Visit 2 <126 mg/dL (<7 mmol/L)
* Hemoglobin A1c (HbA1c) level <6.5%
* Participant willing to use acceptable method of contraception during the study, including the 14-day follow-up period

Exclusion criteria:

* History of malignancy ≤5 years prior to signing informed consent, except for adequately-treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Participation in a study with an investigational compound (non-lipid-modifying) within 30 days
* Pregnant, breastfeeding, or expecting to conceive, or father a child during the study, including the 14-day follow-up period
* Consumption of more than 3 alcoholic drinks on any given day or more than 14 drinks per week
* Engages in or plans to engage in vigorous exercise or an aggressive diet regimen during the study
* Diabetes mellitus, based on medical history, FSG ≥126 mg/dL (7 mmol/L), and HbA1c ≥6.5%
* Risk factors for coronary heart disease
* Active or chronic hepatobiliary or hepatic disease
* Active peptic ulcer disease within 3 months of Visit 1
* History of hypersensitivity or allergic reaction to niacin or niacin-containing products
* Episode of gout within 1 year of Visit 1, unless currently stable on allopurinol
* Taking an LMT (including statins, bile acid sequestrants, fibrates and niacin >50 mg as monotherapy or coadministered with other LMTs)
* Use of over-the- counter or traditional medicine (e.g. red yeast rice products) for lipid-lowering
* Receiving treatment with systemic corticosteroids (unless on stable therapy for at lest 6 weeks for replacement for pituitary/adrenal/hypogonadal disease)
* Uncontrolled illness or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at 37 centers in 2 countries (29 sites in India and 8 sites in Philippines).
Groups:
- ERN/LPRT: Extended-release niacin 1 g in combination with laropiprant 20 mg administered orally once daily for 4 weeks, followed by ERN 2 g LPRT 40 mg administered orally once daily for 12 weeks, to South and Southeast Asian participants with low HDL-C and low-to-moderate coronary heart disease risk.
- Placebo: Matching placebo to ERN/LRPT administered orally once daily for 16 weeks to South and Southeast Asian participants with low HDL-C and low-to-moderate coronary heart disease risk.
Period: Overall Study
Arm/Group | ERN/LPRT | Placebo
Started | 122 | 122
Treated | 120 | 121
Completed | 31 | 39
Not Completed | 91 | 83
Not completed — Adverse Event | 10 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Non-compliance with study drug | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Study terminated by Sponsor | 68 | 75
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERN/LPRT | Placebo | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (9.30) | 45.3 (10.18) | 45.5 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 79 | 172
  Male | 29 | 43 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) Averaged Across Week 12 and Week 16
Description: The percentage change from baseline in the participants' LDL-C was to be evaluated and averaged across treatment Week 12 and Week 16.
Time Frame: Baseline and Weeks 12 to 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in the Ratio of LDL-C to High-Desity Lipoprotein Cholesterol (HDL-C) at Week 16
Description: The percentage from baseline in the participants' ration of LDL-C to HDL-C was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 16
Description: The percentage change from baseline in the participants' HDL-C was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 16
Description: The percentage change from baseline in participants' TG level was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 16
Description: The percentage change from baseline in participants' non-HDL-C was to be calculated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in the Ratio of Total Cholesterol (TC) to HDL-C at Week 16
Description: The percentage change from baseline in the ratio of TC to HDL-C was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) (LP[a]) at Week 16
Description: The pecentage change from baseline in participants LP(a) was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 16
Description: The percentage change from baseline in participants' Apo B was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I (Apo A-I) at Week 16
Description: The percentage change from baseline in participants' Apo A-I was to be evaluated at study Week 16.
Time Frame: Baseline and Week 16
Population: Due to early study termination, this efficacy endpoint was not analyzed.
Arm/Group | ERN/LPRT | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 20 for Serious Adverse Events; Up to Week 18 for Non-Serious Adverse Events.
Description: The safety population consisted of all participants that received at least one dose of study drug.
Arm/Group | ERN/LPRT | Placebo
Serious Adverse Events (participants affected / at risk) | 1/120 | 0/121
Other Adverse Events (participants affected / at risk) | 42/120 | 17/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERN/LPRT (N=120) | Placebo (N=121)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERN/LPRT (N=120) | Placebo (N=121)
Pyrexia (General disorders) | 10 (10) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 7 (7)
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 7 (8) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (25) | 4 (4)
Flushing (Vascular disorders) | 12 (18) | 3 (11)

LIMITATIONS AND CAVEATS:
Due to the small number of participants completing the study (n=70), the resulting underpowered nature of any analyses that might be conducted, and the fact that data are not going to be used, no efficacy analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.